CLINICAL TRIAL: NCT00265278
Title: Double-Blind, Placebo-Controlled Assessment of Interactions Between Intravenous Methamphetamine and Modafinil
Brief Title: Assessment of Interactions Between Intravenous Methamphetamine and Modafinil - 1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-CPU-0008-1
Record Dates: First submitted 2005-12-13; First posted 2005-12-14 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2005-12

CONDITIONS: Amphetamine-Related Disorders
MeSH Terms: conditions — Amphetamine-Related Disorders | interventions — Modafinil

INTERVENTIONS:
Drug: Modafinil

SUMMARY:
The purpose of this study is to assess the potential interactions between intravenous methamphetamine and oral Modafinil.

DETAILED DESCRIPTION:
The primary aims of this experiment are to determine if there are significant safety interactions between oral modafinil and intravenous methamphetamine. Safety will be assessed by measuring adverse events and cardiovascular responses of heart rate (HR), blood pressure (BP), and electrocardiogram (ECG) and stroke distance (ICG).

ELIGIBILITY:
Inclusion Criteria:

* normotensive
* good physical and mental health
* body mass index between 18 and 30
* if female, using an acceptable method of contraception and are not pregnant
* able to give voluntary informed consent

Exclusion Criteria:

* Please contact site for further details

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16
Dates: Start 2005-03; Study Completion 2006-03

PRIMARY OUTCOMES:
Cardiovascular
Subjective symptoms/Mood Effects

CONTACTS AND LOCATIONS:
Overall Officials: Reese Jones, M.D., Principal Investigator — Langley Porter Psychiatric Institute
Locations (1):
- U of CA, San Francisco, San Francisco, California, United States